CLINICAL TRIAL: NCT01435330
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Explore the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Parenterally Administered BVS857 in Healthy Subjects Without and With Insulin Resistance
Brief Title: Safety and Tolerability of BVS857 in Subjects With Insulin Resistance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CBVS857X2101
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Insulin Resistance
Keywords: Safety; BVS857; insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BVS857 (Experimental)
  Interventions: Drug: BVS857
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BVS857
  Arms: BVS857
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will assess the safety, tolerability, drug label and effect in subjects with and without insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects with insulin resistance
* Subjects with controlled hypertension and hyperlipidemia

Exclusion Criteria:

* Smokers
* History of drug or alcohol use
* Autonomic dysfunction
* Significant illness or cardiovascular disease
* Immunodeficiency disease

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Continuously up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Chula Vista, California
  - Novartis Investigative Site, Tacoma, Washington